CLINICAL TRIAL: NCT00705445
Title: Prospective Cluster Randomized Controlled Evaluation of the Impact of Zinc and / or Micronutrient Supplementation on Intestinal Flora, Diarrheal Disease Burden, Intestinal Mucosal Integrity and Growth Among Cohorts of Children in Pakistan
Brief Title: Evaluation of Zinc and / or Micronutrient Supplementation on Intestinal Flora, Diarrheal Disease Burden, Intestinal Mucosal Integrity and Growth Among Children of Pakistan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Dr Zulfiqar Ahmed Bhutta, Professor and Founding Chair, Division of Women and Child Health, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 752-Peds/ERC-07
Record Dates: First submitted 2008-06-25; First posted 2008-06-26 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Malnutrition; Diarrhea; Pneumonia; Growth
Keywords: Malnutrition; Diarrhea; Pneumonia; Growth; Zinc Supplements; Microbiome
MeSH Terms: conditions — Malnutrition; Diarrhea; Pneumonia | interventions — Zinc; Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): This group will not receive any of the intervention supplements. The group will only receive nutritional counselling and education, and treatment provided for any encountered illness according to IMCI guidelines.
  Interventions: Other: Nutritional Counselling and Education
- B (Experimental): This group will receive micronutrient supplements containing microencapsulated Iron, Vitamin C, Vitamin A, Vitamin D, and Folic Acid.
  This group will also receive Nutritional Counselling and Education and treatment according to IMCI Guidelines for any serious illness.
  Interventions: Dietary Supplement: Micronutrient Supplementation without Zinc
- C (Experimental): This group will receive Micronutrient Supplements containing Microencapsulated Iron, Vitamin C, Vitamin A, Vitamin D, Folic Acid, and Zinc.
  This group will also receive nutritional counselling, education and treatment according to IMCI Guidelines in case of any untoward illness.
  Interventions: Dietary Supplement: Micronutrient Supplementation with Zinc

INTERVENTIONS:
Dietary Supplement: Micronutrient Supplementation without Zinc — This will contain Micronutrient Supplements containing Microencapsulated Iron, Vitamin C, Vitamin A, Vitamin D and Folic Acid
  Arms: B
Dietary Supplement: Micronutrient Supplementation with Zinc — This will contain Microencapsulated Iron, Vitamin C, Vitamin A, Vitamin D, and Folic Acid. Additionally, this will also contain 10 mg elemental Zinc Sulphate.
  Arms: C
Other: Nutritional Counselling and Education — This will contain Nutritional Counselling and Education.
  Arms: A

SUMMARY:
Information on the mechanisms of zinc is still in developing phase. Ecological and biological implications of long term zinc supplementation at population level requires assessment. The trial aims to assess the impact of routine supplementation of zinc among young growing children and evaluate its impact on intestinal microbial flora and relationship with gut mucosa integrity and co-morbidities.

DETAILED DESCRIPTION:
WHO has recommended the use of zinc for the treatment of acute diarrhea. Literature supports up-scaling of zinc supplementation programs to prevent childhood illnesses, such as diarrhea and respiratory infections, and its subsequent co-morbid conditions. As the potential mechanisms of action of zinc still remains to be established, this trial is proposed to evaluate the relationship of intestinal microbial flora, intestinal permeability, morbidity patterns and response to various enteric pathogens in a representative birth cohort randomly allocated to receive daily zinc and micronutrients from 6-18 months of age, and a control population.

ELIGIBILITY:
Inclusion Criteria:

* Children of ages 2 weeks to 6 months for recruitment into the Trial. Children of ages 6 months and onwards would eligible to receive intervention (in the form of Micronutrient Sprinkles)

Exclusion Criteria:

* Children with obvious congenital anomalies.

Ages: 2 Weeks to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2745 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Episodes of Diarrhea and additional morbidity such as acute lower respiratory tract infection, pneumonia and days with severe illness. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zulfiqar ZB Bhutta, MBBS, PhD, Principal Investigator — Aga Khan University
Locations (2):
- Pakistan (2):
  - The Aga Khan University, Karachi, Sindh
  - Project Office, Matiari, Matiari, Sindh

REFERENCES:
- [Derived] Balaji V, Dinh DM, Kane AV, Soofi S, Ahmed I, Rizvi A, Chatterjee M, Babji S, Duara J, Moy J, Naumova EN, Wanke CA, Ward HD, Bhutta ZA. Longitudinal Analysis of the Intestinal Microbiota among a Cohort of Children in Rural and Urban Areas of Pakistan. Nutrients. 2023 Feb 28;15(5):1213. doi: 10.3390/nu15051213. PMID 36904212
- [Derived] Popovic A, Bourdon C, Wang PW, Guttman DS, Soofi S, Bhutta ZA, Bandsma RHJ, Parkinson J, Pell LG. Micronutrient supplements can promote disruptive protozoan and fungal communities in the developing infant gut. Nat Commun. 2021 Nov 18;12(1):6729. doi: 10.1038/s41467-021-27010-3. PMID 34795270
- [Derived] Ariff S, Krebs NF, Soofi S, Westcott J, Bhatti Z, Tabassum F, Bhutta ZA. Absorbed zinc and exchangeable zinc pool size are greater in Pakistani infants receiving traditional complementary foods with zinc-fortified micronutrient powder. J Nutr. 2014 Jan;144(1):20-6. doi: 10.3945/jn.113.178715. Epub 2013 Nov 13. PMID 24225451
- [Derived] Soofi S, Cousens S, Iqbal SP, Akhund T, Khan J, Ahmed I, Zaidi AK, Bhutta ZA. Effect of provision of daily zinc and iron with several micronutrients on growth and morbidity among young children in Pakistan: a cluster-randomised trial. Lancet. 2013 Jul 6;382(9886):29-40. doi: 10.1016/S0140-6736(13)60437-7. Epub 2013 Apr 18. PMID 23602230